CLINICAL TRIAL: NCT03810599
Title: Patient-reported Outcomes in the Bergen Early Cardiac Rehabilitation Study
Acronym: BECARES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014/333
Record Dates: First submitted 2018-12-21; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac rehabilitation adherence; Patient-reported outcomes; Post-traumatic growth; Anxiety; Depression; Adherence; Lifestyle; Self-reported health
MeSH Terms: conditions — Coronary Artery Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Pre-post comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early cardiac rehabilitation (Other): Single Group: 5 week cardiac rehabilitation programme. Pre-post comparison.
  Interventions: Other: Early cardiac rehabilitation

INTERVENTIONS:
Other: Early cardiac rehabilitation — This is an early cardiac rehabilitation programme starting 1-2 weeks after hospital discharge (Phase 2A rehabilitation). The programme provided by a multidisciplinary team includes individual counseling, educational sessions and discussion in groups, and exercise training sessions three days a week for five weeks.
  For additional analysis there will be a comparison group that did not receive the intervention for practical reasons.

SUMMARY:
An intervention study with longitudinal follow-up of patients with coronary artery disease undergoing early cardiac rehabilitation is designed.

DETAILED DESCRIPTION:
The main objective of the study is to investigate patient-reported outcomes, their relation to clinical characteristics of the patients and the potential to predict health outcomes and adverse events in coronary artery disease patients participating in an early cardiac rehabilitation programme.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of coronary artery disease
* >=18 years of age
* Has performed a negative exercise test (bike or treadmill) and thereby able to participate in exercise training.

Exclusion Criteria:

* Cognitive impairment
* Unstable angina pectoris
* Aortic stenosis
* Left ventricular ejection fraction <30%
* Heart failure NYHA class III-IV
* Serious arrhythmia in need of treatment
* Being on the waiting list for percutaneous coronary intervention or coronary artery bypass grafting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2013-09-09 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Time to composite of total mortality, and hospitalization for heart failure and atherothrombotic disease (including non-fatal MI, unstable angina and stroke). | Up to 10 years
  Time to combined endpoint from inclusion.

SECONDARY OUTCOMES:
Change in Self-reported health | Immediately after the 5 week intervention, and at 9, 31, 57 and 109 weeks
  The EuroQol 5-dimensions-5 level questionnaire (EQ-5D-5L) is an 5 item self-report-questionnaire assessing self-reported health. The respondent rates each item on a 5-point scale ranging from 1(indicating no problem) to 5 (indicating extreme problems). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change in self-reported global health | Immediately after the 5 week intervention, and at 9, 31, 57 and 109 weeks
  The VAS scale from the EQ-5D-5L assess global health. The scale goes from 0 to 100 were lower score indicates worse health.
Change in post traumatic growth | Immediately after the 5 week intervention, and at 9, 31, 57 and 109 weeks
  The Posttraumatic Growth Inventory-Short Form (PTGI-SF) is a 10 item scale measuring post traumatic growth. The respondent rates each item on a 6-point scale ranging from 0 (I did not experience this change as a result of my crisis) to 5 (I experienced this change to a very great degree as a result of my crisis). The scale is scored by adding all the responses.Individual factors are scored by adding responses to items on each factor. Factors are indicated by the Roman numerals after each item.
Nicotine dependence | Immediately after the 5 week intervention, and at 9, 31, 57 and 109 weeks
  The Fagerström test
Change in anxiety and depression | Immediately after the 5 week intervention, and at 9, 31, 57 and 109 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale where seven of the items relate to anxiety and seven relate to depression. The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence). The total score is 42 (21 per subscale).
Change in physical and mental dimensions of health | Immediately after the 5 week intervention, and at 9, 31, 57 and 109 weeks
  The Short Form Health Survey (SF-12) include 12 items with 3 to 5 response levels. It generates two health indices: mental health and physical health. The score range between 0 and 100, with 100 representing the highest level of health
Change in health status following myocardial infarction | Immediately after the 5 week intervention, and at 9, 31, 57 and 109 weeks
  The Myocardial Infarction Dimensional Assessment Scale (MIDAS) is a PRO measure developed and validated to specifically measure the health status of individuals who have suffered a myocardial infarction. It consist of 7 domains, and is a 35 item scale where respondents rate each item on a 5-point scale ranging from 1 (never) to 5 (always). The function of the MIDAS is to indicate the extent of ill health in each of the seven domains assessed, therefore each dimension is scored separately using a simple scoring methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Tone M Norekvål, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://helse-bergen.no/en/procard/projects-in-procard/patient-reported-outcomes-in-the-bergen-early-cardiac-rehabilitation-study-becarespro